CLINICAL TRIAL: NCT02039479
Title: Randomized, Placebo-controlled Multicenter Trial of Lithium Plus Treatment as Usual (TAU) for Acute Suicidal Ideation and Behavior in Patients With Suicidal Major Depressive Episode
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01KG1307
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Suicidal Ideation/Behavior; Depression
Keywords: anti-suicide; Lithium; Depression; suicidal Ideation/behavior
MeSH Terms: conditions — Suicidal Ideation; Behavior; Depression | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAU + Placebo (Placebo Comparator): Treatment as Usual + Placebo
  Interventions: Drug: Placebo
- TAU + Lithium (Active Comparator): Treatment as Usual + Lithium
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium as Add on to every necessary treatment as usual
  Arms: TAU + Lithium
Drug: Placebo — Placebo as ADD-on to every necessary treatment as usual
  Arms: TAU + Placebo

SUMMARY:
The primary hypothesis of this confirmatory study is that lithium therapy will acutely decrease suicidal ideation and/or suicidal behaviour in inpatients with a major depressive episode (MDE, unipolar and bipolar disorder according to DSM IV criteria). The specific aim is to test the hypothesis that lithium plus treatment as usual (TAU), compared to placebo plus TAU, results in a significantly greater decrease in suicidal ideation and/or behaviour over 5 weeks in inpatients with MDE.

DETAILED DESCRIPTION:
The study will consist of 254 adult patients, hospitalized for a major depressive episode with suicidal ideation and/or behaviour who will be randomized to two groups of each 127 participants. All study participants will receive treatment as usual in the hospital, including (psycho)pharmacological treatment and, if needed, psychotherapy plus a 5-week course of lithium or placebo. Rating scales will be used daily resp. weekly to measure suicidal ideation and/or behaviour, depression, anxiety, mixed/manic features and impulsiveness. Experienced clinicians will rate suicidal ideation and/or behaviour as well as depression twice a week and anxiety, mixed/manic features and impulsiveness once a week.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode; inpatient at screening visit; suicidal ideation/behaviour present defined by a clinical rating of 8 on the Sheehan Suicidality Tracking Scale (S-STS) and a rating of ≥20 on the Montgomery Asberg Depression Scale (MADRS) at both screening and baseline visits; both gender, age 18 years.

Exclusion Criteria:

* Contraindication for and history of lithium treatment within the past 6 months; patient unable to tolerate lithium treatment in the past; comorbid borderline/antisocial personality disorder, currently active substance dependency; patients with acute or unstable severe medical conditions, patients unable to understand the informed consent or involuntary inpatients, positive toxicology screen (illegal drugs), pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
S-STS | 5 Weeks
  Change in the clinician administered (S-STS=Sheehan Suicidality Tracking Scale) total score between initial and final visit

SECONDARY OUTCOMES:
C-SSRS | 5 weeks
  Change of the total score of C-SSRS (Columbia-Suicide Severity Rating Scale) between start and final visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bauer, Prof., Principal Investigator — Dept. of Psychiatry and Psychotherapy; TU Dresden; Ute Lewitzka, MD, Study Director — Dept. of Psychiatry and Psychotherapy, TU Dresden
Locations (5):
- Germany (5):
  - Dept. of Psychiatry and Psychotherapy, Hospital of Dresden Neustadt, Dresden, Saxony
  - Psychiatrie, Verhaltensmedizin und Psychosomatik, Chemnitz
  - Klinik für Psychiatrie, Psychosomatik und Psychotherapie Universitätsklinikum Frankfurt, Frankfurt am Main
  - Psychatrie Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Heidelberg, Heidelberg

REFERENCES:
- [Derived] Lewitzka U, Jabs B, Fulle M, Holthoff V, Juckel G, Uhl I, Kittel-Schneider S, Reif A, Reif-Leonhard C, Gruber O, Djawid B, Goodday S, Haussmann R, Pfennig A, Ritter P, Conell J, Severus E, Bauer M. Does lithium reduce acute suicidal ideation and behavior? A protocol for a randomized, placebo-controlled multicenter trial of lithium plus Treatment As Usual (TAU) in patients with suicidal major depressive episode. BMC Psychiatry. 2015 May 19;15:117. doi: 10.1186/s12888-015-0499-5. PMID 25986590